CLINICAL TRIAL: NCT04785794
Title: Phase 1b Clinical Study to Investigate the Safety and Immunogenicity of the Sing2016 (A/Singapore/INFIMH-16-0019/2016) M2SR H3N2 Monovalent Influenza Vaccine in Adults Ages 50 to 85 Years Old.
Brief Title: Safety and Immunogenicity of the Sing2016 M2SR H3N2 Monovalent Influenza Vaccine in Adults Ages 50 to 85 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FluGen Inc (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FLUGEN-H3N2-V005; DMID 20-0025 (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Three Cohorts will be enrolled sequentially with safety data reviewed between enrollment of successive cohorts.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- M2SR dose, 50-64 years of age (Experimental): Intranasal M2SR vaccine followed by standard, licensed IIV
  Interventions: Biological: Sing2016 M2SR H3N2 influenza vaccine
- Placebo dose, 50-64 years of age (Placebo Comparator): Intranasal physiological saline followed by standard, licensed IIV
  Interventions: Other: Placebo
- M2SR dose, 65-85 years of age (Experimental): Intranasal M2SR vaccine followed by licensed IIV recommended for people 65 years and older
  Interventions: Biological: Sing2016 M2SR H3N2 influenza vaccine
- Placebo dose, 65-85 years of age (Placebo Comparator): Intranasal physiological saline followed by licensed IIV recommended for people 65 years and older
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Sing2016 M2SR H3N2 influenza vaccine — This group will receive a dose of the Sing2016 M2SR H3N2 monovalent influenza vaccine administered intranasally on Day 1 followed by IIV at least 28 days later.
  Arms: M2SR dose, 50-64 years of age; M2SR dose, 65-85 years of age
Other: Placebo — This group will receive saline placebo administered intranasally on Day 1 followed by IIV at least 28 days later.
  Arms: Placebo dose, 50-64 years of age; Placebo dose, 65-85 years of age

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase 1b study to evaluate safety and immunogenicity of the investigational Sing2016 M2SR H3N2 influenza vaccine delivered intranasally to a healthy adult population age 50 to 85 years.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase 1b study to evaluate safety and immunogenicity of the investigational Sing2016 M2SR H3N2 influenza vaccine delivered intranasally to a healthy adult population age 50 to 85 years. Eligible subjects will be randomized 2:1 to receive one administration of Sing2016 M2SR or placebo followed by a dose of age-appropriate licensed inactivated influenza vaccine (IIV) at least 28 days later. Two lead-in groups of adults ages 50-64 years (Cohort 1) and 65 - 85 years (Cohort 2) will be followed by enrollment of an expansion group, ages 65 - 85 (Cohort 3). Safety data will be reviewed between enrollment of successive cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing and able to provide written informed consent.
2. Cohort 1: age 50-64 years at time of enrollment; Cohorts 2 and 3: age 65 to 85 years at time of enrollment (signing of informed consent form).
3. Subject willing to adhere to the requirements of the study and willing and able to communicate with the Investigator and understand the requirements of the study
4. Healthy adults and those with stable chronic conditions as determined by medical history, physical examination, vital signs, clinical safety laboratory examinations and clinical judgment of the investigator to be eligible for study inclusion.
5. Women of child-bearing potential must agree to abstain from sexual intercourse or to correctly use an acceptable method of contraception from 30 days prior to vaccination until 30 days after the last study vaccination.
6. Women of childbearing potential must have a negative urine pregnancy test within 24 hours prior to vaccination with investigational product.

Exclusion Criteria:

1. Any acute or chronic physical or mental condition that would limit the subject's ability to complete the study, increase risk of study participation or participant, or may interfere with interpretation of study results as based on the assessment by the Investigator.
2. Acute or chronic medical condition or history of a medical condition that, in the opinion of the Investigator, would render the study procedures unsafe or would interfere with the evaluation of the responses.
3. Abnormal screening hematology or chemistry value per the FDA Guidance: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials.
4. Currently receiving, or planned to receive during the study, any immunosuppressive therapy.
5. Had a flu-like illness, influenza treatment, influenza vaccination, or prophylactic influenza viral drug administered in the previous 6 months before investigational product administration.
6. Females who are pregnant or nursing; non-vasectomized males, with female partners of child-bearing potential, who are unwilling to use a highly effective form of contraception from the time of enrollment through at least 28 after administration of the investigational product.
7. History of receipt of any investigational vaccine within 28 days of visit 1 or investigational drug within the past six months. An exception is made for receipt of a Covid-19 vaccine whether licensed or under emergency use authorization (EUA) as long as the second dose was given at least 28 days prior to dosing with investigational vaccine.
8. Acute febrile illness within 72 hours prior to investigational product vaccination
9. Receipt of blood/plasma products or immunoglobulin within 6 months before administration of the investigational product or planned for during the period of study participation.
10. Planned donation of blood or blood product of at least approximately 1 pint within 3 months after investigational product administration.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamuk Bilsel, Study Director — FluGen Inc
Locations (3):
- United States (3):
  - Anaheim Clinical Trials, Anaheim, California
  - Accel Clinical, DeLand, Florida
  - Johnson County Clin Trials, Lenexa, Kansas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cohort 1 included subjects ages 50-64 years as a safety check prior to age-escalating to older adults. Cohort 2 included a lead-in group of subjects 65-85 years as a safety check prior to enrolling the expansion group, Cohort 3, in the same age range. Cohorts 2 and 3 received the same treatments and results are combined for these subjects.
Period: Overall Study
Arm/Group | M2SR Dose, 50-64 Years of Age | Placebo Dose, 50-64 Years of Age | M2SR Dose, 65-85 Years of Age | Placebo Dose, 65-85 Years of Age
Started | 10 | 5 | 70 | 37
Completed | 9 | 5 | 67 | 37
Not Completed | 1 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Within each cohort, subjects were to be stratified based on a prescreening antibody titer to HA (by hemagglutinin inhibition [HAI] assay) from Sing2016 H3N2 influenza virus. Subjects were stratified into groups that had a pre-dose HAI titer of <40 and an HAI titer from 40 to <320.
Groups:
- Total: Total of all reporting groups
Arm/Group | M2SR Dose, 50-64 Years of Age | Placebo Dose, 50-64 Years of Age | M2SR Dose, 65-85 Years of Age | Placebo Dose, 65-85 Years of Age | Total
Number analyzed (Participants) | 10 | 5 | 70 | 37 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 5 | 0 | 0 | 15
  >=65 years | 0 | 0 | 70 | 37 | 107
Age, Continuous [Median (Standard Deviation); unit: years] | 57 (3.1) | 57 (2.9) | 70 (4.2) | 73 (4.6) | 72 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 46 | 23 | 78
  Male | 5 | 1 | 24 | 14 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 8 | 2 | 10
  Not Hispanic or Latino | 10 | 5 | 62 | 35 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 7 | 1 | 8
  White | 10 | 5 | 61 | 34 | 110
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 70 | 37 | 122
Baseline HAI titer to A/Sing2016 [Count of Participants; unit: Participants]
  <40 | 8 | 3 | 34 | 18 | 63
  40 to <=320 | 2 | 2 | 36 | 19 | 59

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent AEs During 7 Days After Experimental Treatment
Description: The number and percentage of study participants who experience local (at the dose administration site) and systemic (throughout the body) reactions during the 7 days after administration of investigational M2SR vaccine or placebo. Solicited and unsolicited signs and symptoms were reported as AEs after review by the Investigator or designee, either separately using the corresponding Medical Dictionary for Regulatory Activities (MedDRA) terminology of the sign or symptom or combined using the appropriate term.
Time Frame: Day 1 to Day 8
Population: All subjects who received an IP dose
Measure: Count of Participants; unit: Participants
Arm/Group | M2SR Dose, 50-64 Years of Age | Placebo Dose, 50-64 Years of Age | M2SR Dose, 65-85 Years of Age | Placebo Dose, 65-85 Years of Age
Number analyzed (Participants) | 10 | 5 | 70 | 37
Participants | 1 | 0 | 12 | 3

2. Primary Outcome: Treatment Emergent AEs During 28 Days After Experimental Treatment
Description: The number and percentage of study participants who experience a treatment emergent AE during the 28 days after administration of investigational M2SR vaccine or placebo. Unsolicited signs and symptoms were reported as AEs after review by the Investigator or designee, either separately using the corresponding MedDRA terminology of the sign or symptom or combined using the appropriate term.
Time Frame: Day 1 to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | M2SR Dose, 50-64 Years of Age | Placebo Dose, 50-64 Years of Age | M2SR Dose, 65-85 Years of Age | Placebo Dose, 65-85 Years of Age
Number analyzed (Participants) | 10 | 5 | 70 | 37
Participants | 1 | 1 | 16 | 8

3. Primary Outcome: SAEs Through 28 Days After Licensed IIV Treatment
Description: The number and percentage of study participants who experience SAEs from the time of study entry through 28 days after receipt of IIV. Unsolicited signs and symptoms were reported as AEs after review by the Investigator or designee, either separately using the corresponding MedDRA terminology of the sign or symptom or combined using the appropriate term.
Time Frame: Time of enrollment through 28 days after receipt of IIV where the IIV was administered an average of 49 days post-IP and with an interval up to 91 days later.
Population: Numbers of subjects analyzed for SAEs includes 2 subjects who were administered IIV but who did not have biological samples collected and therefore were not considered to have completed trial. Thus, the participant flow shows 9 subjects completed while safety shows 10 subjects for the M2SR dose 50-64 years of age. Similarly, the participant flow shows 67 subjects completed while safety shows 68 subjects for the M2SR dose 65-85 years of age.
Measure: Count of Participants; unit: Participants
Arm/Group | M2SR Dose, 50-64 Years of Age | Placebo Dose, 50-64 Years of Age | M2SR Dose, 65-85 Years of Age | Placebo Dose, 65-85 Years of Age
Number analyzed (Participants) | 10 | 5 | 68 | 37
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: IP administration until 28 days post-IIV (where interval between IP and IIV was up to 91 days with an average span of 49 days)
Description: Includes treatment emergent AEs
Arm/Group | M2SR Dose, 50-64 Years of Age | Placebo Dose, 50-64 Years of Age | M2SR Dose, 65-85 Years of Age | Placebo Dose, 65-85 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/70 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 0/70 | 0/37
Other Adverse Events (participants affected / at risk) | 1/10 | 1/5 | 2/70 | 3/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | M2SR Dose, 50-64 Years of Age (N=10) | Placebo Dose, 50-64 Years of Age (N=5) | M2SR Dose, 65-85 Years of Age (N=70) | Placebo Dose, 65-85 Years of Age (N=37)
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
headache (Nervous system disorders) | 0 | 0 | 1 | 2
muscle strain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the results of the Study will be made in conjunction with the presentation of a joint, multicenter publication of the Study results with the investigators and the institutions from all appropriate sites contributing data. If such a multicenter publication is not submitted within 24 months after conclusion of the Study at all sites, then Investigator may publish the results from their Site individually,

DOCUMENTS (2):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT04785794/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT04785794/SAP_001.pdf